CLINICAL TRIAL: NCT06381024
Title: A Study of the Benefit of Telemonitoring for Hospital Staff Treating Patients With Oral or Intravenous Cancer Treatments: a French Prospective, Randomized, Unblinded, Single-centre Study.
Brief Title: A Study of Telemonitoring in Cancer Patients
Acronym: MINERVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Bligny (Other)
Collaborators: Exystat (Other); Cureety (Industry); Pharmaspecific (Unknown); ProPens (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022 A02702-41
Record Dates: First submitted 2024-02-28; First posted 2024-04-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: remote patient monitoring
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients initiating either oral or intravenous chemotherapy for cancer will be randomly allocated in a 1:1 ratio to either:
  * In-person care alone (Standard of care group).
  * In-person care with telemonitoring (Standard of care with Cureety group).
  The randomization will be stratified by:
  • Oral versus intravenous cancer treatment. The number of patients initiating oral treatment at randomization will be restricted to 20 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care group (No Intervention): Standard of care
- Standard of care with Cureety group (Experimental): In-person care with remote patient monitoring with the Cureety application
  Interventions: Device: remote patient monitoring

INTERVENTIONS:
Device: remote patient monitoring — Cureety is a digital telemonitoring platform, specifically designed to monitor signs and symptoms of disease progression and AEs in cancer patients. The digital tool is adaptable to specific treatments and disease settings. The platform collects various data including treatment delays, dose reductions, quality of life and safety data. In terms of safety, once configured for the treatment and disease setting, the patient responds to an electronic PRO (ePRO) questionnaire based on the NCI-CTCAE version (v)5.0.10 Depending on the responses, an algorithm classifies patients as either "correct", "compromised", "state to be monitored", or "critical state". Depending on the classification, patients are notified of the actions to be taken.
  Other Names: Cureety
  Arms: Standard of care with Cureety group

SUMMARY:
The goal of this prospective, randomized, unblinded, single-centre, interventional study is to assess the effectiveness of standard of care with Cureety, compared to standard of care alone, to reduce the number of all telephone calls during the first 4 months of oral or intravenous cancer treatment for patients older than 18 years of age, initiating oral or intravenous cancer treatment at the Centre Hospitalier de Bligny.

Patients initiating either oral or intravenous chemotherapy for cancer will be randomly allocated in a 1:1 ratio to either:

* In-person care alone (Standard of care group).
* In-person care with Cureety telemonitoring (Standard of care with Cureety group).

Participants will:

* be monitored with digital application Cureety (Standard of care with Cureety group)
* fill out quality of life questionnaire (baseline, 2 months, 4 months)
* fill out satisfaction questionnaire (2 months, 4 months)
* have the ongoing and incoming phone calls logged (duration and type)

DETAILED DESCRIPTION:
Rationale:

Telemonitoring of cancer patients provides patients with cancer-related information, as well as allowing appointment management, early detection of side-effects/adverse events (AEs), and the collection of safety and quality of life data from the patients' perspectives.1 Several studies have assessed the benefit of telemonitoring from the patients' perspective.1-5 However, few studies have investigated the benefit of telemonitoring for healthcare professionals.4,6,7 The Symptom Tracking and Reporting (STAR) randomized trial, performed at the Memorial Sloan Kettering Institute, randomly allocated patients to either usual care or the patient-reported outcome (PRO) group.8,9 Patients in the PRO group completed a web-based questionnaire concerning 12 common AEs (based on the National Cancer Institute Common Terminology Criteria for AEs [NCI-CTCAE version (v) 5.0]10) at or between visits. In the PRO group, 63% of patients reported severe AEs during the study. Patients, in the PRO group, reported improved quality of life, fewer admissions to emergency rooms or hospitalization, extended duration of chemotherapy, and extended overall survival (OS). This increased OS is potentially due to the early response by healthcare professionals to severe AEs identified by the web-based questionnaire. For healthcare professionals, the study reported fewer unscheduled visits for patients allocated to the PRO group.

Interestingly, in the STAR trial, 77% of the nurse interventions (either by email or telephone) were in response to alerts (either counseling or symptom management), 12% were for initiating or changing of supportive treatment, 8% were for referrals to the emergency room or hospital, 2% were for chemotherapy dose modifications, and 2% were for ordering imagery or biological test.11 In France, the Foch hospital initiated the Star program for patients undergoing chemotherapy.12 The program collects patient data within at most 3 days prior to each chemotherapy session and transfer these to healthcare professionals to prepare the chemotherapy. The patient has the choice of completing a questionnaire via the internet or providing the information by telephone with the aid of a nurse. The data includes health status, presence of AEs, and blood test results. These data allow healthcare professionals to adapt or delay the chemotherapy, change treatments, and provide the patient with personalized advice according to the patient's health status. The program has improved the performance of departments involved by increasing the number of patients treated per day, decreasing the waiting times for patients, and by reducing the wastage of healthcare products.

Consequently, numerous French healthcare centers want to implement programs like the Star program. However, a substantial portion of the data collection occurs via the telephone, particularly outgoing calls (from the hospital staff to patients). This increase in telephone communication means more work for healthcare professions. A digital telemonitoring platform, like Cureety that can collect this data before chemotherapy, is expected to decrease outgoing calls by between 30% to 50% and facilitate the implementing of these programs.

Furthermore, healthcare centers in France are continually facing budget restrictions. At the same time, treating cancer patients is associated with an increase in incoming calls from patients during cancer treatment, particularly for minor AEs. The treating of these incoming calls is often repetitive and time consuming for hospital staff. The collection of data concerning AEs, of varying severity, can be integrated in a digital platform. Patients with minor AEs can be provided with the actions to be followed via the platform. This will allow staff to concentrate on patients with severe AEs needing urgent attention.

Cureety is a digital telemonitoring platform, specifically designed to monitor signs and symptoms of disease progression and AEs in cancer patients. The digital tool is adaptable to specific treatments and disease settings. The platform collects various data including treatment delays, dose reductions, quality of life and safety data. In terms of safety, once configured for the treatment and disease setting, the patient responds to an electronic PRO (ePRO) questionnaire based on the NCI-CTCAE version (v)5.0.10 Depending on the responses, an algorithm classifies patients as either "correct", "compromised", "state to be monitored", or "critical state". Depending on the classification, patients are notified of the actions to be taken.

This study will assess the benefit of adding Cureety telemonitoring to standard of care, compared to standard of care alone, for monitoring cancer patients undergoing oral or intravenous cancer treatments.

Methodology:

The MINERVA study was designed as a prospective, randomized, unblinded, single-centre, interventional study with minimal risks and constraints for patients.

Patients initiating either oral or intravenous chemotherapy for cancer will be randomly allocated in a 1:1 ratio to either:

* In-person care alone (Standard of care group).
* In-person care with telemonitoring (Standard of care with Cureety group).

The randomization will be stratified by:

• Oral versus intravenous cancer treatment. The number of patients initiating oral treatment at randomization will be restricted to 20 patients.

Data concerning the telephone calls between study patients and the staff at the CH Bligny will be collected. The incoming and outgoing calls from the CH Bligny will be classified in the following categories:

* Cancer treatments information (including the use of associated prophylactic treatments, e.g., granulocyte colony-stimulating factor [G-CSF], antihistamines etc.)
* Appointments, in the following subcategories:

  * Administration of cancer therapy (including oral and intravenous treatments, etc.).
  * Consultations for a reason other than administering therapy.
  * Blood tests and other examinations.
* Prescriptions.
* Biological examinations (in preparation for cancer treatment).
* Psychological support.
* Patient education and supportive care.
* Cancer treatment-related AEs.
* Non-cancer treatment-related AEs, excluding COVID-related.
* COVID-related.
* Related to Cureety.
* Other calls. The planned enrolment period is 5 months. The planned follow-up period for each patient is 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that have provide written informed consent for study participation.
2. Patients aged 18 years or older.
3. Patients initiating oral or intravenous treatment (chemotherapy, immunotherapy, targeted therapies etc.) for localized or metastatic or recurrent cancer treated at the CH Bligny.
4. Patients with the capacity, personally (e.g., language and capacity to use the application), and in terms of infrastructure (internet access, possessing a smart phone etc.) to perform telemonitoring with Cureety.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2

Exclusion Criteria:

* Patients treated for cancer at the CH Bligny in the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Number of all telephone calls during the first 4 months of oral or intravenous cancer treatment | 4 months after randomization
  Number of calls, defined as the number of incoming and outgoing calls that occurs during the 4 months from randomization

SECONDARY OUTCOMES:
Duration of all telephone calls during the first 4 months of oral or intravenous cancer treatment | During 4 months after randomization
Numbers of telephone calls during the first 4 months of cancer treatment in subgroups | During 4 months after randomization
  Numbers of telephone calls during the first 4 months of cancer treatment in subgroups: Incoming calls, Outgoing calls, categories of calls
Hospital-free survival rate | During 4 months after randomization
  Hospital-free survival (HFS) is defined as the time interval (in days) without any hospitalization from randomization until death of any cause.
Quality of life at 2 and 4 months after initiation of cancer treatment. | During 4 months after randomization
  Quality of life (QoL) in the study groups will be compared using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire14 measured relative to baseline at 2 and 4 months (±3 weeks) after randomization. The QoL will be compared overall and according to the scales
Patient satisfaction with the healthcare provided | During 4 months after randomization
  Patient satisfaction with the healthcare provided, in the study groups, will be compared using 4-point Likert scale (1 for not at all satisfied to 4 completely satisfied), measured at 2 and 4 months (±3 weeks) after randomization.
CH Bligny staff satisfaction with the healthcare provided | At 12 months after first inclusion
  • CH Bligny staff satisfaction with the healthcare provided, in the study groups, will be compared using a specific questionnaire provided to the staff at the end of the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Bligny, Briis-sous-Forges, France

IPD SHARING:
Plan to Share IPD: No